CLINICAL TRIAL: NCT02593721
Title: Hypoalgesic Effect of Median Nerve Neural Mobilization Versus Ibuprofen Pharmacologic Treatment in Patients With Cervicobrachial Pain
Brief Title: Hypoalgesic Effect of Neural Mobilization Versus Ibuprofen Pharmacologic Treatment
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Francisco Unda Solano, PHD Student, Universidad Europea de Madrid
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CE0072015
Record Dates: First submitted 2015-10-26; First posted 2015-11-02 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Cervicobrachial Neuralgia
MeSH Terms: conditions — Brachial Plexus Neuritis | interventions — Ibuprofen; Midol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Median Nerve Neural Mobilization (Experimental): 15 minute Median Nerve Neural Mobilization sessions 5 times a week (monday to Friday) during 6 continuous weeks The maximum degree of elbow extension applied in the Median Nerve neural mobilization procedure was determined through the use of a Universal Goniometer Device.
  Interventions: Procedure: Median Nerve Neural Mobilization
- Ibuprofen (Active Comparator): A single daily 400 mg dose of oral Ibuprofen that can be increased depending on patient tolerance to a maximum dose of 1200 mg/day equally divided in 3 oral intakes of the drug every 8 hours during 6 continuous weeks.
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Procedure: Median Nerve Neural Mobilization — Non-surgical non-invasive Median Nerve neural mobilization procedure was applied by a physical therapist continuously during 2 minutes in 5 different occasions with 1 minute of rest between each 2 minute application of the Neural Mobilization technique. The intervention was applied during a period of 6 weeks. The maximum level of elbow extension movement degree without the reproduction of symptoms during the application of the Median Nerve Neural mobilization treatment was determined through the baseline use of a Universal Goniometer Device.
  Other Names: Neural Tissue Mobilization of the Median Nerve; Median Nerve Neurodynamics
  Arms: Median Nerve Neural Mobilization
Drug: Ibuprofen — The active comparator group received an oral Ibuprofen treatment. The starting dose was of 400 mg/day and it was increased to a maximum of 1200 mg/day divided in 3 oral intakes every 8 hours depending on patient tolerance.The intervention was applied during a period of 6 weeks.
  Other Names: Addaprin®; Advil®; Caldolor®; Cedaprin®; I-Prin®; Midol®; Motrin®; Motrin® IB; NeoProfen®; Profen IB®; Proprinal®; Ultraprin®
  Arms: Ibuprofen

SUMMARY:
The purpose of this study is to compare the effectivity of Median Nerve Neural Mobilization and oral Ibuprofen in treating patients who suffer cervicobrachial pain

DETAILED DESCRIPTION:
Median Nerve Neural Mobilization and Ibuprofen both relieve cervicobrachial pain, but this happens through different mechanisms and with a different onset of side effects. Median Nerve Neural Mobilization is a physical therapy technique that achieves pain relief through mechanical stimulation of the median nerve and the brachial plexus. The proper mechanical stimulation of the nerve and its surrounding neural tissue induces a wide variety of physiologic responses that may reduce cervicobrachial pain including the activation of descending nervous system pain modulation mechanisms, all though the entire set of underlying reasons for this pain reduction is not completely understood. Among the effects caused by the Neural Tissue Mobilization that produce pain relief are: intraneural edema reduction, changes on the intraneural nerve pressure,dispersion of pro-inflammatory substances and an increase in nerve mobility

Ibuprofen is a nonsteroidal anti-inflammatory drug used worldwide to control pain, fever and inflammation.Oral intake of Ibuprofen produces a hypoalgesic effect due to biochemical inhibition of the COX enzymes, which convert arachidonic acid to prostaglandin H2 (PGH2). PGH2, which in turn, is converted by other enzymes to several types of prostaglandins and thromboxanes (which are mediators of pain and inflammation).

Side effects derived from the oral intake of Ibuprofen are related to its systemic action and can be severe in some patients. This fact suggests that oral Ibuprofen may not be suitable to use in all types of patients suffering from cervicobrachial pain, meanwhile the Median Nerve Neural Mobilization has little to no side effects known. This reveals a point of interest in determining comparative effectiveness between this two therapeutic options in the treatment of cervicobrachial pain.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of cervicobrachial pain confirmed by magnetic resonance imaging
* Presence of unilateral symptoms of arm pain, paresthesia or numbness in the upper extremity during at least 3 continuous months previous to the application of treatment.
* Positive results in all of the following tests: Spurling, Distraction, and Upper Limb

Exclusion Criteria:

* Contraindication in the use of nonsteroidal anti inflammatory drugs (NSAIDs)
* The use of any type of treatment, therapy, procedure or drug to relieve pain
* Patients who are under anticonvulsant, antidepressant or psychotropic medication
* Vertebral instability
* Vertebral osteoporosis
* Vertebral or spine infection.
* Neurologic diseases of genetic, infectious or neoplastic origin
* Cervical stenosis myelopathy
* Pregnancy
* Kinesiophobia
* Endocrine disorders and menopause
* History of spine surgery
* Intellectual disability, severe mental illness, intoxication, severe sleep deprivation, Alzheimer's disease.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2015-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline using the Numeric Rating Scale for Pain at 1 hour | at baseline and 1 hour after the application of treatment, corresponding to intervention sessions 1, 15 and 30
  The Numeric Rating Scale (NRS) is an 11 point scale for patient self-reporting of pain, it was employed to evaluate the presence and relieve of cervicobrachial pain symptoms

SECONDARY OUTCOMES:
Change from baseline of the Physical function involving the affected upper limb using the Quik DASH Scale | at baseline, corresponding to intervention session 1 and 30 of treatment.
  The Disabilities of the Arm, Shoulder and Hand ( QuickDASH) Test is a self-report short questionnaire designed to measure physical function and symptoms in people with any of several musculoskeletal disorders of the upper limb.
Change from baseline cervical rotation range of motion at 1 hour | at baseline and 1 hour after the application of treatment, corresponding to intervention sessions 1 and 30
  Cervical rotation was assessed in units of rotation degrees, using the cervical range-of-motion device (CROM).

CONTACTS AND LOCATIONS:
Overall Officials: Francisco H Unda, PT, MSc, Principal Investigator — Universidad Europea de Madrid
Locations (1):
- Centro de Medicina Fisica y de Rehabilitacion FISIOREH, Valencia, Carabobo, Venezuela

REFERENCES:
- [Result] Cowell IM, Phillips DR. Effectiveness of manipulative physiotherapy for the treatment of a neurogenic cervicobrachial pain syndrome: a single case study -- experimental design. Man Ther. 2002 Feb;7(1):31-8. doi: 10.1054/math.2001.0429. PMID 11884154
- [Result] Salt E, Wright C, Kelly S, Dean A. A systematic literature review on the effectiveness of non-invasive therapy for cervicobrachial pain. Man Ther. 2011 Feb;16(1):53-65. doi: 10.1016/j.math.2010.09.005. Epub 2010 Nov 12. PMID 21075037
- [Result] Allison GT, Nagy BM, Hall T. A randomized clinical trial of manual therapy for cervico-brachial pain syndrome -- a pilot study. Man Ther. 2002 May;7(2):95-102. doi: 10.1054/math.2002.0453. PMID 12151246
- [Result] Huisstede BM, Bierma-Zeinstra SM, Koes BW, Verhaar JA. Incidence and prevalence of upper-extremity musculoskeletal disorders. A systematic appraisal of the literature. BMC Musculoskelet Disord. 2006 Jan 31;7:7. doi: 10.1186/1471-2474-7-7. PMID 16448572
- [Result] Radhakrishnan K, Litchy WJ, O'Fallon WM, Kurland LT. Epidemiology of cervical radiculopathy. A population-based study from Rochester, Minnesota, 1976 through 1990. Brain. 1994 Apr;117 ( Pt 2):325-35. doi: 10.1093/brain/117.2.325. PMID 8186959
- [Result] Daffner SD, Hilibrand AS, Hanscom BS, Brislin BT, Vaccaro AR, Albert TJ. Impact of neck and arm pain on overall health status. Spine (Phila Pa 1976). 2003 Sep 1;28(17):2030-5. doi: 10.1097/01.BRS.0000083325.27357.39. PMID 12973155
- [Result] Isabel de-la-Llave-Rincon A, Puentedura EJ, Fernandez-de-Las-Penas C. Clinical presentation and manual therapy for upper quadrant musculoskeletal conditions. J Man Manip Ther. 2011 Nov;19(4):201-11. doi: 10.1179/106698111X13129729551985. PMID 23115473
- [Result] Antonelli BA, de Paula Xavier AA, Oenning P, Baumer MH, da Silva TF, Pilatti LA. Prevalence of cervicobrachial discomforts in elementary school teachers. Work. 2012;41 Suppl 1:5709-14. doi: 10.3233/WOR-2012-0927-5709. PMID 22317661
- [Result] Dillingham TR. Evaluating the patient with suspected radiculopathy. PM R. 2013 May;5(5 Suppl):S41-9. doi: 10.1016/j.pmrj.2013.03.015. Epub 2013 Mar 19. PMID 23524070
- [Result] Boyles R, Toy P, Mellon J Jr, Hayes M, Hammer B. Effectiveness of manual physical therapy in the treatment of cervical radiculopathy: a systematic review. J Man Manip Ther. 2011 Aug;19(3):135-42. doi: 10.1179/2042618611Y.0000000011. PMID 22851876
- [Result] Eubanks JD. Cervical radiculopathy: nonoperative management of neck pain and radicular symptoms. Am Fam Physician. 2010 Jan 1;81(1):33-40. PMID 20052961
- [Result] Peolsson A, Soderlund A, Engquist M, Lind B, Lofgren H, Vavruch L, Holtz A, Winstrom-Christersson A, Isaksson I, Oberg B. Physical function outcome in cervical radiculopathy patients after physiotherapy alone compared with anterior surgery followed by physiotherapy: a prospective randomized study with a 2-year follow-up. Spine (Phila Pa 1976). 2013 Feb 15;38(4):300-7. doi: 10.1097/BRS.0b013e31826d2cbb. PMID 23407407
- [Result] Caridi JM, Pumberger M, Hughes AP. Cervical radiculopathy: a review. HSS J. 2011 Oct;7(3):265-72. doi: 10.1007/s11420-011-9218-z. Epub 2011 Sep 9. PMID 23024624
- [Result] Young IA, Michener LA, Cleland JA, Aguilera AJ, Snyder AR. Manual therapy, exercise, and traction for patients with cervical radiculopathy: a randomized clinical trial. Phys Ther. 2009 Jul;89(7):632-42. doi: 10.2522/ptj.20080283. Epub 2009 May 21. PMID 19465371
- [Result] Campbell WW. Evaluation and management of peripheral nerve injury. Clin Neurophysiol. 2008 Sep;119(9):1951-65. doi: 10.1016/j.clinph.2008.03.018. Epub 2008 May 14. PMID 18482862
- [Result] Walton Walter WJ. Brain´s Diseases Of The Nervous System. London: Oxford UP; 1969.
- [Result] Nikolaidis I, Fouyas IP, Sandercock PA, Statham PF. Surgery for cervical radiculopathy or myelopathy. Cochrane Database Syst Rev. 2010 Jan 20;2010(1):CD001466. doi: 10.1002/14651858.CD001466.pub3. PMID 20091520
- [Result] Legakis A, Boyd BS. The influence of scapular depression on upper limb neurodynamic test responses. J Man Manip Ther. 2012 May;20(2):75-82. doi: 10.1179/2042618611Y.0000000020. PMID 23633886
- [Result] McGregor AH, Probyn K, Cro S, Dore CJ, Burton AK, Balague F, Pincus T, Fairbank J. Rehabilitation following surgery for lumbar spinal stenosis. Cochrane Database Syst Rev. 2013 Dec 9;2013(12):CD009644. doi: 10.1002/14651858.CD009644.pub2. PMID 24323844
- [Result] Cleland JA, Whitman JM, Fritz JM, Palmer JA. Manual physical therapy, cervical traction, and strengthening exercises in patients with cervical radiculopathy: a case series. J Orthop Sports Phys Ther. 2005 Dec;35(12):802-11. doi: 10.2519/jospt.2005.35.12.802. PMID 16848101
- [Result] Beneciuk JM, Bishop MD, George SZ. Effects of upper extremity neural mobilization on thermal pain sensitivity: a sham-controlled study in asymptomatic participants. J Orthop Sports Phys Ther. 2009 Jun;39(6):428-38. doi: 10.2519/jospt.2009.2954. PMID 19487826
- [Result] Elvey R HT. Neural tissue evaluation and treatment, Donatelli R, Physical Therapy of the Shoulder,. 3rd ed. Livingstone C, editor. New York; 1997
- [Result] Fritz JM, Thackeray A, Brennan GP, Childs JD. Exercise only, exercise with mechanical traction, or exercise with over-door traction for patients with cervical radiculopathy, with or without consideration of status on a previously described subgrouping rule: a randomized clinical trial. J Orthop Sports Phys Ther. 2014 Feb;44(2):45-57. doi: 10.2519/jospt.2014.5065. Epub 2014 Jan 9. PMID 24405257
- [Result] Persson LC, Carlsson CA, Carlsson JY. Long-lasting cervical radicular pain managed with surgery, physiotherapy, or a cervical collar. A prospective, randomized study. Spine (Phila Pa 1976). 1997 Apr 1;22(7):751-8. doi: 10.1097/00007632-199704010-00007. PMID 9106315
- [Result] Carlesso LC, Macdermid JC, Gross AR, Walton DM, Santaguida PL. Treatment preferences amongst physical therapists and chiropractors for the management of neck pain: results of an international survey. Chiropr Man Therap. 2014 Mar 24;22(1):11. doi: 10.1186/2045-709X-22-11. PMID 24661461
- [Result] Coppieters MW, Stappaerts KH, Wouters LL, Janssens K. The immediate effects of a cervical lateral glide treatment technique in patients with neurogenic cervicobrachial pain. J Orthop Sports Phys Ther. 2003 Jul;33(7):369-78. doi: 10.2519/jospt.2003.33.7.369. PMID 12918862
- [Result] Garland EL. Treating chronic pain: the need for non-opioid options. Expert Rev Clin Pharmacol. 2014 Sep;7(5):545-50. doi: 10.1586/17512433.2014.928587. Epub 2014 Jun 11. PMID 24918159
- [Result] Santos FM, Grecco LH, Pereira MG, Oliveira ME, Rocha PA, Silva JT, Martins DO, Miyabara EH, Chacur M. The neural mobilization technique modulates the expression of endogenous opioids in the periaqueductal gray and improves muscle strength and mobility in rats with neuropathic pain. Behav Brain Funct. 2014 May 13;10:19. doi: 10.1186/1744-9081-10-19. PMID 24884961
- [Result] Ogneva IV. Cell mechanosensitivity: mechanical properties and interaction with gravitational field. Biomed Res Int. 2013;2013:598461. doi: 10.1155/2013/598461. Epub 2012 Dec 26. PMID 23509748
- [Result] Bonin RP, Bories C, De Koninck Y. A simplified up-down method (SUDO) for measuring mechanical nociception in rodents using von Frey filaments. Mol Pain. 2014 Apr 16;10:26. doi: 10.1186/1744-8069-10-26. PMID 24739328
- [Result] Moriarty O, Finn DP. Cognition and pain. Curr Opin Support Palliat Care. 2014 Jun;8(2):130-6. doi: 10.1097/SPC.0000000000000054. PMID 24722475
- [Result] Woolf CJ. Central sensitization: implications for the diagnosis and treatment of pain. Pain. 2011 Mar;152(3 Suppl):S2-S15. doi: 10.1016/j.pain.2010.09.030. Epub 2010 Oct 18. PMID 20961685
- [Result] Courtney CA, Clark JD, Duncombe AM, O'Hearn MA. Clinical presentation and manual therapy for lower quadrant musculoskeletal conditions. J Man Manip Ther. 2011 Nov;19(4):212-22. doi: 10.1179/106698111X13129729552029. PMID 23115474
- [Result] Woolf CJ, Salter MW. Neuronal plasticity: increasing the gain in pain. Science. 2000 Jun 9;288(5472):1765-9. doi: 10.1126/science.288.5472.1765. PMID 10846153
- [Result] Woolf CJ. Central sensitization: uncovering the relation between pain and plasticity. Anesthesiology. 2007 Apr;106(4):864-7. doi: 10.1097/01.anes.0000264769.87038.55. No abstract available. PMID 17413924
- [Result] Santos FM, Silva JT, Giardini AC, Rocha PA, Achermann AP, Alves AS, Britto LR, Chacur M. Neural mobilization reverses behavioral and cellular changes that characterize neuropathic pain in rats. Mol Pain. 2012 Jul 29;8:57. doi: 10.1186/1744-8069-8-57. PMID 22839415
- [Result] Villafane JH. Botulinum toxin type A combined with neurodynamic mobilization for lower limb spasticity: a case report. J Chiropr Med. 2013 Mar;12(1):39-44. doi: 10.1016/j.jcm.2013.01.001. PMID 23997723
- [Result] Villafane JH, Pillastrini P, Borboni A. Manual therapy and neurodynamic mobilization in a patient with peroneal nerve paralysis: a case report. J Chiropr Med. 2013 Sep;12(3):176-81. doi: 10.1016/j.jcm.2013.10.007. PMID 24396318
- [Result] Ellis RF, Hing WA, McNair PJ. Comparison of longitudinal sciatic nerve movement with different mobilization exercises: an in vivo study utilizing ultrasound imaging. J Orthop Sports Phys Ther. 2012 Aug;42(8):667-75. doi: 10.2519/jospt.2012.3854. Epub 2012 Jun 18. PMID 22711174
- [Result] Shacklock M. Neural mobilization: a systematic review of randomized controlled trials with an analysis of therapeutic efficacy. J Man Manip Ther. 2008;16(1):23-4. doi: 10.1179/106698108790818602. No abstract available. PMID 19119381
- [Result] Lin PL, Shih YF, Chen WY, Ma HL. Neurodynamic responses to the femoral slump test in patients with anterior knee pain syndrome. J Orthop Sports Phys Ther. 2014 May;44(5):350-7. doi: 10.2519/jospt.2014.4781. Epub 2014 Apr 14. PMID 24730437
- [Result] Franze K. The mechanical control of nervous system development. Development. 2013 Aug;140(15):3069-77. doi: 10.1242/dev.079145. PMID 23861056
- [Result] Livne A, Bouchbinder E, Geiger B. Cell reorientation under cyclic stretching. Nat Commun. 2014 May 30;5:3938. doi: 10.1038/ncomms4938. PMID 24875391
- [Result] Lopez-Fagundo C, Bar-Kochba E, Livi LL, Hoffman-Kim D, Franck C. Three-dimensional traction forces of Schwann cells on compliant substrates. J R Soc Interface. 2014 Aug 6;11(97):20140247. doi: 10.1098/rsif.2014.0247. PMID 24872498
- [Result] Nee RJ, Vicenzino B, Jull GA, Cleland JA, Coppieters MW. Neural tissue management provides immediate clinically relevant benefits without harmful effects for patients with nerve-related neck and arm pain: a randomised trial. J Physiother. 2012;58(1):23-31. doi: 10.1016/S1836-9553(12)70069-3. PMID 22341379
- [Result] Savva C, Giakas G. The effect of cervical traction combined with neural mobilization on pain and disability in cervical radiculopathy. A case report. Man Ther. 2013 Oct;18(5):443-6. doi: 10.1016/j.math.2012.06.012. Epub 2012 Jul 18. PMID 22818658
- [Result] Ellis RF, Hing WA. Neural mobilization: a systematic review of randomized controlled trials with an analysis of therapeutic efficacy. J Man Manip Ther. 2008;16(1):8-22. doi: 10.1179/106698108790818594. PMID 19119380
- [Result] van der Velde G, Hogg-Johnson S, Bayoumi AM, Cassidy JD, Cote P, Boyle E, Llewellyn-Thomas H, Chan S, Subrata P, Hoving JL, Hurwitz E, Bombardier C, Krahn M. Identifying the best treatment among common nonsurgical neck pain treatments: a decision analysis. J Manipulative Physiol Ther. 2009 Feb;32(2 Suppl):S209-18. doi: 10.1016/j.jmpt.2008.11.021. PMID 19251067
- [Result] Sheather-Reid RB, Cohen M. Efficacy of analgesics in chronic pain: a series of N-of-1 studies. J Pain Symptom Manage. 1998 Apr;15(4):244-52. doi: 10.1016/s0885-3924(98)00369-8. PMID 9601160
- [Result] Nemes D, Amaricai E, Tanase D, Popa D, Catan L, Andrei D. Physical therapy vs. medical treatment of musculoskeletal disorders in dentistry--a randomised prospective study. Ann Agric Environ Med. 2013;20(2):301-6. PMID 23772581
- [Result] Yamamoto M, Sugano T, Kashiwazaki S, Kageyama T, Mizushima Y, Kameyama M. Double-blind comparison of piroxicam and indomethacin in the treatment of cervicobrachial syndrome and periarthritis scapulohumeralis (stiff shoulder). Eur J Rheumatol Inflamm. 1983;6(3):266-73. PMID 6391931
- [Result] Rainsford KD. Ibuprofen: from invention to an OTC therapeutic mainstay. Int J Clin Pract Suppl. 2013 Jan;(178):9-20. doi: 10.1111/ijcp.12055. PMID 23163543
- [Result] Grace D, Rogers J, Skeith K, Anderson K. Topical diclofenac versus placebo: a double blind, randomized clinical trial in patients with osteoarthritis of the knee. J Rheumatol. 1999 Dec;26(12):2659-63. PMID 10606379
- [Result] Welsch P, Sommer C, Schiltenwolf M, Hauser W. [Opioids in chronic noncancer pain-are opioids superior to nonopioid analgesics? A systematic review and meta-analysis of efficacy, tolerability and safety in randomized head-to-head comparisons of opioids versus nonopioid analgesics of at least four week's duration]. Schmerz. 2015 Feb;29(1):85-95. doi: 10.1007/s00482-014-1436-0. German. PMID 25376546
- [Result] Kuchari E, Han S, Karlowicz-Bodalska K, Miskiewicz K, Kutycka E. Safety of oral ibuprofen--analysis of data from the spontaneous reporting system in Poland. Acta Pol Pharm. 2014 Jul-Aug;71(4):687-90. PMID 25272896
- [Result] World Health Organisation Medicines E. Essential Medicines WHO Model List ( revised March 2005 ) Explanatory Notes. World Heal Organ. 2005;(14).
- [Result] Vyas FI, Rana DA, Patel PM, Patel VJ, Bhavsar RH. Randomized comparative trial of efficacy of paracetamol, ibuprofen and paracetamol-ibuprofen combination for treatment of febrile children. Perspect Clin Res. 2014 Jan;5(1):25-31. doi: 10.4103/2229-3485.124567. PMID 24551584
- [Result] Kanabar D. A practical approach to the treatment of low-risk childhood fever. Drugs R D. 2014 Jun;14(2):45-55. doi: 10.1007/s40268-014-0052-x. PMID 24916274
- [Result] Adatia A, Rainsford KD, Kean WF. Osteoarthritis of the knee and hip. Part II: therapy with ibuprofen and a review of clinical trials. J Pharm Pharmacol. 2012 May;64(5):626-36. doi: 10.1111/j.2042-7158.2012.01456.x. Epub 2012 Feb 7. PMID 22471358
- [Result] Bradley JD, Brandt KD, Katz BP, Kalasinski LA, Ryan SI. Comparison of an antiinflammatory dose of ibuprofen, an analgesic dose of ibuprofen, and acetaminophen in the treatment of patients with osteoarthritis of the knee. N Engl J Med. 1991 Jul 11;325(2):87-91. doi: 10.1056/NEJM199107113250203. PMID 2052056
- [Result] Wagner JG, Albert KS, Szpunar GJ, Lockwood GF. Pharmacokinetics of ibuprofen in man IV: absorption and disposition. J Pharmacokinet Biopharm. 1984 Aug;12(4):381-99. doi: 10.1007/BF01062664. PMID 6527231
- [Result] Hall AH, Smolinske SC, Stover B, Conrad FL, Rumack BH. Ibuprofen overdose in adults. J Toxicol Clin Toxicol. 1992;30(1):23-37. doi: 10.3109/15563659208994443. PMID 1542147
- [Result] Auriel E, Regev K, Korczyn AD. Nonsteroidal anti-inflammatory drugs exposure and the central nervous system. Handb Clin Neurol. 2014;119:577-84. doi: 10.1016/B978-0-7020-4086-3.00038-2. PMID 24365321
- [Result] Volans G, Monaghan J, Colbridge M. Ibuprofen overdose. Int J Clin Pract Suppl. 2003 Apr;(135):54-60. PMID 12723749
- [Result] Rodriguez SC, Olguin AM, Miralles CP, Viladrich PF. Characteristics of meningitis caused by Ibuprofen: report of 2 cases with recurrent episodes and review of the literature. Medicine (Baltimore). 2006 Jul;85(4):214-220. doi: 10.1097/01.md.0000229757.78057.50. PMID 16862046
- [Result] Bancos S, Bernard MP, Topham DJ, Phipps RP. Ibuprofen and other widely used non-steroidal anti-inflammatory drugs inhibit antibody production in human cells. Cell Immunol. 2009;258(1):18-28. doi: 10.1016/j.cellimm.2009.03.007. Epub 2009 Apr 5. PMID 19345936
- [Result] Imani F, Motavaf M, Safari S, Alavian SM. The therapeutic use of analgesics in patients with liver cirrhosis: a literature review and evidence-based recommendations. Hepat Mon. 2014 Oct 11;14(10):e23539. doi: 10.5812/hepatmon.23539. eCollection 2014 Oct. PMID 25477978
- [Result] Moriarty O, McGuire BE, Finn DP. The effect of pain on cognitive function: a review of clinical and preclinical research. Prog Neurobiol. 2011 Mar;93(3):385-404. doi: 10.1016/j.pneurobio.2011.01.002. Epub 2011 Jan 7. PMID 21216272
- [Result] Asghar W, Jamali F. The effect of COX-2-selective meloxicam on the myocardial, vascular and renal risks: a systematic review. Inflammopharmacology. 2015 Feb;23(1):1-16. doi: 10.1007/s10787-014-0225-9. Epub 2014 Dec 17. PMID 25515365
- [Result] Krenkel O, Mossanen JC, Tacke F. Immune mechanisms in acetaminophen-induced acute liver failure. Hepatobiliary Surg Nutr. 2014 Dec;3(6):331-43. doi: 10.3978/j.issn.2304-3881.2014.11.01. PMID 25568858
- [Result] Rasu RS, Vouthy K, Crowl AN, Stegeman AE, Fikru B, Bawa WA, Knell ME. Cost of pain medication to treat adult patients with nonmalignant chronic pain in the United States. J Manag Care Spec Pharm. 2014 Sep;20(9):921-8. doi: 10.18553/jmcp.2014.20.9.921. PMID 25166291
- [Result] Orlando BJ, Lucido MJ, Malkowski MG. The structure of ibuprofen bound to cyclooxygenase-2. J Struct Biol. 2015 Jan;189(1):62-6. doi: 10.1016/j.jsb.2014.11.005. Epub 2014 Nov 25. PMID 25463020
- [Result] O'Rielly DD, Loomis CW. Increased expression of cyclooxygenase and nitric oxide isoforms, and exaggerated sensitivity to prostaglandin E2, in the rat lumbar spinal cord 3 days after L5-L6 spinal nerve ligation. Anesthesiology. 2006 Feb;104(2):328-37. doi: 10.1097/00000542-200602000-00019. PMID 16436853
- [Result] Forster C, Magerl W, Beck A, Geisslinger G, Gall T, Brune K, Handwerker HO. Differential effects of dipyrone, ibuprofen, and paracetamol on experimentally induced pain in man. Agents Actions. 1992 Jan;35(1-2):112-21. doi: 10.1007/BF01990960. PMID 1509971
- [Result] Litalien C, Jacqz-Aigrain E. Risks and benefits of nonsteroidal anti-inflammatory drugs in children: a comparison with paracetamol. Paediatr Drugs. 2001;3(11):817-58. doi: 10.2165/00128072-200103110-00004. PMID 11735667
- [Result] Borenstein D. Low Back and Neck Pain. Low Back and Neck Pain [Internet]. 2004. p. 771-849.
- [Result] Sniezek PJ, Brodland DG, Zitelli JA. A randomized controlled trial comparing acetaminophen, acetaminophen and ibuprofen, and acetaminophen and codeine for postoperative pain relief after Mohs surgery and cutaneous reconstruction. Dermatol Surg. 2011 Jul;37(7):1007-13. doi: 10.1111/j.1524-4725.2011.02022.x. Epub 2011 May 11. PMID 21561527
- [Result] Jeyakumar A, Brickman TM, Williamson ME, Hirose K, Krakovitz P, Whittemore K, Discolo C. Nonsteroidal anti-inflammatory drugs and postoperative bleeding following adenotonsillectomy in pediatric patients. Arch Otolaryngol Head Neck Surg. 2008 Jan;134(1):24-7. doi: 10.1001/archoto.2007.11. PMID 18209131
- [Result] Moore RA, Derry S, Wiffen PJ, Straube S, Aldington DJ. Overview review: Comparative efficacy of oral ibuprofen and paracetamol (acetaminophen) across acute and chronic pain conditions. Eur J Pain. 2015 Oct;19(9):1213-23. doi: 10.1002/ejp.649. Epub 2014 Dec 22. PMID 25530283
- [Result] Kissin I. Scientometric assessment of drugs for chronic pain, 1979-2013: rapid growth of publications, paucity of successful drugs. J Pain Res. 2014 Aug 20;7:505-14. doi: 10.2147/JPR.S67479. eCollection 2014. PMID 25187736
- [Result] Unzueta A, Vargas HE. Nonsteroidal anti-inflammatory drug-induced hepatoxicity. Clin Liver Dis. 2013 Nov;17(4):643-56, ix. doi: 10.1016/j.cld.2013.07.009. Epub 2013 Sep 4. PMID 24099022
- [Result] Herndon CM, Dankenbring DM. Patient perception and knowledge of acetaminophen in a large family medicine service. J Pain Palliat Care Pharmacother. 2014 Jun;28(2):109-16. doi: 10.3109/15360288.2014.908993. Epub 2014 May 12. PMID 24813653
- [Result] Zadrazil J. [Nonsteroidal antiinflammatory drugs and the kidney]. Vnitr Lek. 2006 Jul-Aug;52(7-8):686-90. Czech. PMID 16967609
- [Result] Waddington F, Naunton M, Thomas J. Paracetamol and analgesic nephropathy: Are you kidneying me? Int Med Case Rep J. 2014 Dec 15;8:1-5. doi: 10.2147/IMCRJ.S71471. eCollection 2015. PMID 25548527
- [Result] Whelton A, Hamilton CW. Nonsteroidal anti-inflammatory drugs: effects on kidney function. J Clin Pharmacol. 1991 Jul;31(7):588-98. doi: 10.1002/j.1552-4604.1991.tb03743.x. PMID 1894754
- [Result] Turajane T, Wongbunnak R, Patcharatrakul T, Ratansumawong K, Poigampetch Y, Songpatanasilp T. Gastrointestinal and cardiovascular risk of non-selective NSAIDs and COX-2 inhibitors in elderly patients with knee osteoarthritis. J Med Assoc Thai. 2009 Dec;92 Suppl 6:S19-26. PMID 20128070
- [Result] van der Linden MW, van der Bij S, Welsing P, Kuipers EJ, Herings RM. The balance between severe cardiovascular and gastrointestinal events among users of selective and non-selective non-steroidal anti-inflammatory drugs. Ann Rheum Dis. 2009 May;68(5):668-73. doi: 10.1136/ard.2007.087254. Epub 2008 May 21. PMID 18495734
- [Result] Ingrasciotta Y, Sultana J, Giorgianni F, Caputi AP, Arcoraci V, Tari DU, Linguiti C, Perrotta M, Nucita A, Pellegrini F, Fontana A, Cavagna L, Santoro D, Trifiro G. The burden of nephrotoxic drug prescriptions in patients with chronic kidney disease: a retrospective population-based study in Southern Italy. PLoS One. 2014 Feb 18;9(2):e89072. doi: 10.1371/journal.pone.0089072. eCollection 2014. PMID 24558471
- [Result] Chaparro LE, Wiffen PJ, Moore RA, Gilron I. Combination pharmacotherapy for the treatment of neuropathic pain in adults. Cochrane Database Syst Rev. 2012 Jul 11;2012(7):CD008943. doi: 10.1002/14651858.CD008943.pub2. PMID 22786518
- [Result] Cohen SP, Hayek S, Semenov Y, Pasquina PF, White RL, Veizi E, Huang JH, Kurihara C, Zhao Z, Guthmiller KB, Griffith SR, Verdun AV, Giampetro DM, Vorobeychik Y. Epidural steroid injections, conservative treatment, or combination treatment for cervical radicular pain: a multicenter, randomized, comparative-effectiveness study. Anesthesiology. 2014 Nov;121(5):1045-55. doi: 10.1097/ALN.0000000000000409. PMID 25335172
- [Result] Schmid A, Brunner F, Wright A, Bachmann LM. Paradigm shift in manual therapy? Evidence for a central nervous system component in the response to passive cervical joint mobilisation. Man Ther. 2008 Oct;13(5):387-96. doi: 10.1016/j.math.2007.12.007. Epub 2008 Mar 3. PMID 18316238
- [Result] Harvey MP, Descarreaux M. Short term modulation of trunk neuromuscular responses following spinal manipulation: a control group study. BMC Musculoskelet Disord. 2013 Mar 13;14:92. doi: 10.1186/1471-2474-14-92. PMID 23496876
- [Result] McReynolds TM, Sheridan BJ. Intramuscular ketorolac versus osteopathic manipulative treatment in the management of acute neck pain in the emergency department: a randomized clinical trial. J Am Osteopath Assoc. 2005 Feb;105(2):57-68. PMID 15784928
- [Result] Dabbs V, Lauretti WJ. A risk assessment of cervical manipulation vs. NSAIDs for the treatment of neck pain. J Manipulative Physiol Ther. 1995 Oct;18(8):530-6. PMID 8583176
- [Result] Vicenzino B, Collins D, Benson H, Wright A. An investigation of the interrelationship between manipulative therapy-induced hypoalgesia and sympathoexcitation. J Manipulative Physiol Ther. 1998 Sep;21(7):448-53. PMID 9777544
- [Result] Bahreini M, Jalili M, Moradi-Lakeh M. A comparison of three self-report pain scales in adults with acute pain. J Emerg Med. 2015 Jan;48(1):10-8. doi: 10.1016/j.jemermed.2014.07.039. Epub 2014 Sep 27. PMID 25271179
- [Result] Arumugam V, Selvam S, MacDermid JC. Radial nerve mobilization reduces lateral elbow pain and provides short-term relief in computer users. Open Orthop J. 2014 Oct 17;8:368-71. doi: 10.2174/1874325001408010368. eCollection 2014. PMID 25352930
- [Result] Price DD, Bush FM, Long S, Harkins SW. A comparison of pain measurement characteristics of mechanical visual analogue and simple numerical rating scales. Pain. 1994 Feb;56(2):217-226. doi: 10.1016/0304-3959(94)90097-3. PMID 8008411
- [Result] Youdas JW, Carey JR, Garrett TR. Reliability of measurements of cervical spine range of motion--comparison of three methods. Phys Ther. 1991 Feb;71(2):98-104; discussion 105-6. doi: 10.1093/ptj/71.2.98. PMID 1989013
- [Result] Audette I, Dumas JP, Cote JN, De Serres SJ. Validity and between-day reliability of the cervical range of motion (CROM) device. J Orthop Sports Phys Ther. 2010 May;40(5):318-23. doi: 10.2519/jospt.2010.3180. PMID 20436238
- [Result] Fletcher JP, Bandy WD. Intrarater reliability of CROM measurement of cervical spine active range of motion in persons with and without neck pain. J Orthop Sports Phys Ther. 2008 Oct;38(10):640-5. doi: 10.2519/jospt.2008.2680. PMID 18827326
- [Result] Svensson P, Arendt-Nielsen L, Nielsen H, Larsen JK. Effect of chronic and experimental jaw muscle pain on pain-pressure thresholds and stimulus-response curves. J Orofac Pain. 1995 Fall;9(4):347-56. PMID 8995906
- [Result] Angst F, Schwyzer HK, Aeschlimann A, Simmen BR, Goldhahn J. Measures of adult shoulder function: Disabilities of the Arm, Shoulder, and Hand Questionnaire (DASH) and its short version (QuickDASH), Shoulder Pain and Disability Index (SPADI), American Shoulder and Elbow Surgeons (ASES) Society standardized shoulder assessment form, Constant (Murley) Score (CS), Simple Shoulder Test (SST), Oxford Shoulder Score (OSS), Shoulder Disability Questionnaire (SDQ), and Western Ontario Shoulder Instability Index (WOSI). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S174-88. doi: 10.1002/acr.20630. No abstract available. PMID 22588743
- [Result] Moshe S, Izhaki R, Chodick G, Segal N, Yagev Y, Finestone AS, Juven Y. Predictors of return to work with upper limb disorders. Occup Med (Lond). 2015 Oct;65(7):564-9. doi: 10.1093/occmed/kqv100. Epub 2015 Jul 20. PMID 26195341
- See also: DASH Outcome Measure Institute for Work & Health — http://dash.iwh.on.ca/about-dash